CLINICAL TRIAL: NCT06443918
Title: A Just-in-Time Adaptive Intervention for Child and Family Mental Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colliga Apps Corp. (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R44MH123368 (NIH); R44MH123368 (NIH)
Record Dates: First submitted 2024-02-23; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Mental Health and Well-being; Family Functioning
Keywords: Mental health and well-being; Child development; Digital mental health; Digital intervention; Family functioning
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Half of families will be randomly assigned to the intervention group. The intervention will include family-based activities for improving child and family mental health and functioning delivered as psychoeducation and activities through the smartphone app. The intervention also includes real-time feedback and coaching of family interactions through a just-in-time adaptive intervention (JITAI).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be informed during consent that they will have a 50-50 chance of receiving the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention aims to improve child and family mental health and functioning through psychoeducation and family-based activities delivered via a smartphone app. This intervention also includes a just-in-time adaptive intervention (JITAI) for coaching family interactions in real-time. Caregivers will wear smartwatches and carry smartphones for 8 weeks. Children will wear smartwatches. A variety of types of data will be collected from the phones and watches, such as heart rate, activity levels, and sleep. We will also collect daily surveys, daily audio recordings, a 15-minute survey every 2 weeks about their experiences using the app, and check-in calls every 2 weeks.
  Interventions: Behavioral: A Just-in-Time Adaptive Intervention for Child and Family Mental Health
- Control group (No Intervention): Caregivers will wear smartwatches and carry smartphones for 8 weeks. Children will wear smartwatches. Participants will complete placebo psychoeducational modules matched in length and reading level to the intervention content. A variety of types of data will be collected from the phones and watches, such as heart rate, activity levels, and sleep. We will also collect daily surveys, daily audio recordings, a 15-minute survey every 2 weeks about their experiences using the app, and check-in calls every 2 weeks.

INTERVENTIONS:
Behavioral: A Just-in-Time Adaptive Intervention for Child and Family Mental Health — Families in the intervention group will download an app on their smartphones. The app will deliver psychoeducational modules and family-based homework activities. It will include a component where AI is used to assess the quality of family-based interactions and provide in-the-moment feedback and coaching to guide the family interaction.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to test an app-based just-in-time-adaptive intervention (JITAI). The intervention aims to improve child and family mental health. A JITAI provides in-the-moment feedback to coach families. The questions it tests are if the app will improve mental health and family functioning. Participants will download an app on their phone and complete JITAI sessions. Researchers will compare intervention and control groups to see if the app improves mental health.

DETAILED DESCRIPTION:
The following study tests the efficacy of an app-based program designed to improve child and family mental health and well-being. The intervention will include family-based activities for improving child and family mental health and functioning delivered as psychoeducation and activities through the smartphone app, as well as a just-in-time adaptive intervention (JITAI) component where AI analysis for family interactions will be used to provide real-time, dynamic feedback to families. Participants will be informed during consent that they will have a 50-50 chance of receiving the intervention. The study will assess caregiver and child functioning in a variety of domains, such as mental health symptoms, attachment style, and family conflict through a series of baseline and follow-up questionnaires. Caregivers may use their own smartphones, or they will be lent smartphones for the study. Caregivers and children will also be lent Fitbits/Apple Watches. The intervention will last 8 weeks. Data will include daily surveys, daily audio recordings, 15-minute surveys every 2 weeks about their experiences using the app, bi-weekly check-ins, psychoeducational modules, homework activities, JITAI sessions, and passively sensed data. The intervention will be administered through the smartphone app and will include daily 5-15-minute psychoeducation modules and practice sessions and daily JITAI sessions.

ELIGIBILITY:
Inclusion criteria:

* A family income less than or equal to the 33rd percentile for their county of residence OR
* At least one participating family member identifies as belonging to an ethnic/racial minoritized group AND
* Child mental health symptoms at or above the 70th percentile based on any subscale of the Strengths and Difficulties Questionnaire AND
* Participants speak English and/or Spanish AND
* Have a child 6-9 years old at the time of enrollment AND
* Families must be located in Texas or Florida

Exclusion Criteria:

* Active suicidal ideation OR
* Active homicidal ideation OR
* Current child abuse OR
* Current violence in the home

Families meeting these exclusion criteria will undergo a clinical risk assessment and be referred for alternative treatment services.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 357 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Child mental health symptoms measured by the Child Behavior Checklist | 8 weeks
  Children in the intervention group will evidence decreased mental health symptoms compared to children in the control group.
Child attachment measured via the Attachment Style Classification Questionnaire for Latency Age Children | 8 weeks
  Children in the intervention group will evidence increased secure attachment compared to children in the control group.
Parent-child conflict measured via the Parent-Child Conflict Tactics Scale | 8 weeks
  Children in the intervention group will evidence decreased parent-child conflict compared to children in the control group.

SECONDARY OUTCOMES:
Caregiver mental health measured via the Symptoms Checklist 27-Plus | 8 weeks
  Caregivers in the intervention group will evidence decreased mental health symptoms compared to caregivers in the control group.
Caregiver attachment measured via the Experiences in Close Relationships Scale | 8 weeks
  Caregivers in the intervention group will evidence increased secure attachment compared to caregivers in the control group.
Inter-parental conflict measured via the Conflict Tactics Scale | 8 weeks
  Caregivers in the intervention group will evidence decreased inter-parental conflict compared to caregivers in the control group.

OTHER OUTCOMES:
Child physical health measured via the Child Health Questionnaire | 8 weeks
  Children in the intervention group will evidence decreased physical health symptoms compared to children in the control group.
Caregiver physical health measured via the Patient Health Questionnaire | 8 weeks
  Caregivers in the intervention group will evidence decreased physical health symptoms compared to parents in the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ahle, B.S., Principal Investigator — Colliga Apps; Adela Timmons, Ph.D., Principal Investigator — The University of Texas at Austin; Jonthan Comer, Ph.D., Principal Investigator — Florida International University
Locations (2):
- United States (2):
  - Florida International University, Miami, Florida
  - The University of Texas at Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Researchers can request access to data through Colliga's website by filling out a request form at: https://colliga.io/data-repository/.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available within 1 year after the completion of the clinical trial. Individual requests for data access will be processed within 3 months. Data will be available for individual researchers' use for 1 year with an opportunity to renew yearly. The repository will be maintained for at least 3 years.
Access Criteria: Requests can be submitted by providing the researcher's name, contact information, desired date of dataset access, and explanation for the use of data. Colliga Apps administrators will process requests and give access to approved and verified researchers after the completion of a data use agreement.
URL: https://colliga.io/data-repository/

REFERENCES:
- See also: Colliga Apps website — http://colliga.io